CLINICAL TRIAL: NCT00140946
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Two-Period, Parallel-group Study to Assess the Effect of Montelukast Sodium With Concomitant Administration of Inhaled Budesonide in Asthmatic Patients.
Brief Title: A Study to Assess the Effect of Montelukast Sodium With Concomitant Administration of Inhaled Budesonide in Asthmatic Patients (0476-075)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-075; MK0476-075; 2005_057
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0476; montelukast sodium/Duration of Treatment: 16 weeks
Drug: Comparator: placebo / Duration of Treatment: 16 weeks

SUMMARY:
A study to assess the clinical effect of montelukast sodium with concomitant administration of inhaled budesonide in asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 70 with asthma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 1998-03; Primary Completion 2000-10 (Actual); Study Completion 2000-10 (Actual)

PRIMARY OUTCOMES:
Percentage of days of asthma exacerbations

SECONDARY OUTCOMES:
Percentage of asthma free days
Percentage of nocturnal awakenings
Beta agonist use

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Vaquerizo MJ, Casan P, Castillo J, Perpina M, Sanchis J, Sobradillo V, Valencia A, Verea H, Viejo JL, Villasante C, Gonzalez-Esteban J, Picado C; CASIOPEA (Capacidad de Singulair Oral en la Prevencion de Exacerbaciones Asmaticas) Study Group. Effect of montelukast added to inhaled budesonide on control of mild to moderate asthma. Thorax. 2003 Mar;58(3):204-10. doi: 10.1136/thorax.58.3.204. PMID 12612294